CLINICAL TRIAL: NCT03815955
Title: Reducing Sedentary Behaviour at St. Joseph's Primary Care Diabetes Support Program; Effect on Blood Glucose Levels in Patients With Type II Diabetes
Brief Title: Reducing Sedentary Behaviour in Patients With Type II Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Collaborators: St. Joseph's Health Care London (Other)
Responsible Party: Principal Investigator, Dr. Harry Prapavessis, Principal Investigator, Western University, Canada
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 112907
Record Dates: First submitted 2019-01-18; First posted 2019-01-25 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2; Sedentary Lifestyle
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2; Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-Sedentary Behaviour Group (Experimental): Participants in this arm will model the primary care team as they engage in minimal sedentary behaviour and replace sitting with standing and light, incidental movements.
  Interventions: Behavioral: Non-Sedentary Behaviour Modelling
- Standard Care Control Group (No Intervention): Participants that are limited to standing, due to amputations, diabetic foot pain and ulcers, or sensory diabetic neuropathy, will follow standard care and attend the DIGMA in a seated position.

INTERVENTIONS:
Behavioral: Non-Sedentary Behaviour Modelling — Consistent with social learning theory, the primary care provider and the DIGMA support team will model, demonstrate, and verbalize aspects of increased confidence to perform the 1-hour appointment in a standing position and offer a variety of strategies to cope and overcome any feelings of discomfort. Emphasis will be placed on the strategies the primary care team uses to break sitting with standing and light, incidental movements. It will be anticipated that the participant will observe cues and relevant information specific to their behaviour change and engage in minimal sedentary behaviour.
  Arms: Non-Sedentary Behaviour Group

SUMMARY:
The study will implement a prospective one-arm feasibility study. After an initial eligibility screening by the primary care provider during their intake appointment, new patients will be invited to participate in an acute intervention to reduce sedentary behaviour during a group appointment at St. Joseph's Primary Care Diabetes Support (SJHC PCDSP). Scheduled with up to 10 other people, participants will be encouraged to model the primary care provider and support team as they engage in minimal sedentary behaviour and replace sitting with standing and light, incidental movements.

An accelerometer-based sensory (ActivPAL4) will be worn and used to measure the patients' sedentary behaviour and physical activity patterns, including the duration and frequency of breaks in sedentary time during the appointment. Capillary blood glucose differences will be assessed at pre- and post-appointment. A series of paper-pencil questionnaires will also measure self-efficacy, goal intention, and positive and negative affect at both pre- and post-appointment.

DETAILED DESCRIPTION:
Following pre-screening at their intake appointment, if appropriate for a DIGMA and eligible to participate, new patients to SJHC PCDSP will be invited to attend a DIGMA scheduled two-weeks post-intake appointment. Participants will provide their written informed consent and patient demographic information, assessed by questionnaire, during the first hour of their appointment. With a trained research assistant, the participant will complete a series of behavioural measures including: the Godin Leisure-Time Exercise Questionnaire (GLTEQ) and a modified Sedentary Behaviour Questionnaire (SBQ). Standardized anthropometric measurements, including waist circumference, weight, height, and capillary blood glucose, of all participants will also be completed separately in an exam room.

Consistent with social learning theory, the primary care provider and the DIGMA support team will model, demonstrate, and verbalize aspects of increased confidence to perform the 1-hour appointment in a standing position and offer a variety of strategies to cope and overcome any feelings of discomfort. Emphasis will be placed on the strategies the primary care models uses to break sitting with standing and light, incidental movements. It will be anticipated that the participant will observe cues and relevant information specific to their behaviour change and engage in minimal sedentary behaviour.

The frequency of breaks and the duration of breaks taken during the scheduled DIGMA will be measured using an ActivPAL4 monitor, a wearable device that can measure sitting/lying, standing, and walking time, sit-to-stand and stand-to-sit transition counts and step counts.

Capillary blood glucose will be measured by the research staff at both pre- and post-appointment using a glucometer. As patients are not required to restrict their diet before a standard DIGMA, there will be no restrictions on food and/or drink intake before/during the morning of, the travel to, and/or during the appointment. Participants will be asked to self-report the time and what they ate during their last meal in their demographics questionnaire.

Self-efficacy and positive and negative affect will be self-reported at both pre- and post-appointment using a scale adapted from the General Self-Efficacy Scale and the Positive and Negative Affect Schedule (PANAS), respectively. As well, goal intentions of the patients will be measured using a questionnaire along three dimensions: respondents will refer to a specific point in time, to the place, and to the degree of behavioural intent that is linked to the situational context specified by time and place. An example of one of the questions will be "Over the next week, do you intend to sit less at home?". Subjects will then indicate using a 5-point Likert scale the degree to which they endorse this statement (e.g., 1 is not at all to 5 is completely agree).

ELIGIBILITY:
Inclusion Criteria:

* Participants, aged 18 years or older, will be eligible if they present diagnostic criteria according to the Diabetes Canada 2018 Clinical Practice Guidelines for the Prevention and Management of Diabetes in Canada for type 2 diabetes (diagnosed by any of the following criteria: glycated hemoglobin (A1C) ≥6.5%, fasting plasma glucose (FPG) ≥7.0 mmol/L, 2-hour plasma glucose (2hPG) in a 75 g oral glucose tolerance test (OGTT) ≥11.1 mmol/L, random PG ≥11.1 mmol/L) and would benefit from a DIGMA.

Exclusion Criteria:

* Individuals with diabetes will be excluded if they are younger than 18 years, have significant illness, or an inability to communicate in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-03-14 (Actual); Primary Completion 2019-04-25 (Actual); Study Completion 2019-04-25 (Actual)

PRIMARY OUTCOMES:
Frequency of Non-Sedentary Behaviour Breaks | The ActivPAL4 will be worn during the whole 1-hour DIGMA, and will record the frequency of breaks during this time (60 minutes).
  The frequency of breaks taken from engaging in sedentary behaviour recorded during the scheduled 1-hour appointment with the primary care provider will be measured using the ActivPAL4 monitor, a wearable device specifically designed for sedentary behaviour interventions. The ActivPAL4 can measure sitting/lying, standing, and walking time, sit-to-stand and stand-to-sit transition counts and step counts.
Non-Sedentary Behaviour Break Time | The ActivPAL4 will be worn during the whole 1-hour DIGMA, and will record the duration of breaks during this time (60 minutes).
  The duration of breaks (minutes) taken during the scheduled 1-hour appointment with the primary care provider will be measured using the ActivPAL4 monitor, a wearable device specifically designed for sedentary behaviour interventions. The ActivPAL4 can measure sitting/lying, standing, and walking time, sit-to-stand and stand-to-sit transition counts and step counts.
Capillary Blood Glucose | Capillary blood glucose differences will be assessed at the start of their DIGMA (0 minutes), and will be re-assessed after their appointment (60 minutes).
  Capillary blood glucose (mg/dl) of all participants will be measured by the research staff at both pre- and post-appointment using a Accu-chek Guide meter and test strips (glucometer).
Self-efficacy | Self-efficacy will be self-measured at the start of their DIGMA (0 minutes), and will be re-assessed after their appointment (60 minutes).
  Self-efficacy will be assessed using a scale adapted from the General Self-Efficacy Scale. Participants will rate their confidence to standing for 5 minutes during decreasing periods of time (i.e., +3 hours, 2 hours, 1 hour, <1 hour). An example of one of the statements used will be "I believe that I can stand for 5 minutes every +3hours". Participants will also rate their confidence to standing and moving for increasing periods of time (i.e., 2 minutes, 5 minutes, 10 minutes, and 20 minutes) over a 2-hour time interval. An example of one of the statements used will be "I believe that I can stand and move for 2 minutes ever 2 hours".
Goal Intentions | Goal intentions will be assessed at the start of their DIGMA (0 minutes), and will be re-assessed after their appointment (60 minutes).
  Goal intentions will be measured through the completion of a questionnaire along three dimensions: respondents will refer to a specific point in time, to the place, and to the degree of behavioral intent that is linked to the situational context specified by time and place. An example of one of the statements used will be "Over the next week, I intend to stand more at home". Subjects will then indicate using a 5-point Likert scale the degree to which they endorse this statement (e.g., 1 is not at all to 5 is completely agree).
Positive and Negative Affect | Positive and negative affect will be assessed at the start of their DIGMA (0 minutes), and will be re-assessed after their appointment (60 minutes).
  Positive and negative affect will be self-reported using the 20-item questionnaire, Positive and Negative Affect Schedule (PANAS).

CONTACTS AND LOCATIONS:
Overall Officials: Harry Prapavessis, PhD, Principal Investigator — University of Western Ontario, Canada
Locations (2):
- Canada (2):
  - University of Western Ontario, London, Ontario
  - St. Joseph's Family Medical and Dental Centre, London, Ontario